CLINICAL TRIAL: NCT03456271
Title: A Prospective Cohort Study:Forecast Fracture Risk With a Serum Marker of Type 2 Diabetes in Guangzhou Community
Status: Terminated | Type: Observational
Why Stopped: limited Patient recruitment
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-NFMDXK-001
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes Mellitus and Fragility Fractures
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fracture group
- non-fracture group

INTERVENTIONS:
Other:

SUMMARY:
The objective of this study is to find out the biochemical markers which have independent predictive value of fragility fractures risk with Type 2 diabetes in Guangzhou community and evaluate bone strength better and increase the ability of recognizing fracture risk through following-up visits the bone metabolism index like esRAGE-to-pentosidine ratio of the petients with type 2 diabetes and osteoporosis,compared with the classical fracture risk assessment instrument.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18-65 years; (2) patients were diagnosed with type 2 diabetes based on the definition of diabetes of WHO in 1999.

Exclusion Criteria:

* 1. type 1 diabetes and other specific types of diabetes; 2. diabetes related acute complications like diabetic ketoacidosis and hyperglycemic hyperosmolar status. 3. had used drugs that is known to have effect on bone(like active vitamin D, bisphosphonate, calcitonin, estrogen receptor modulators, estrogen, thiazolidinediones); 4. suffer from diseases that is known to have effect on bone (hyperthyroidism, hypothyroidism, hyperparathyroidism, hypoparathyroidism,cushing syndrome,chronic renal failure,renal tubular acidosis,osteoporosis after gastrectomy,osteoporosis caused by liver disease,rheumatoid disease,osteoporosis induced by gastrointestinal absorption dysfunction); 5. disuse osteoporosis; 6. cannot be exposure to sunlight due to skin diseases; 7. use glucocorticoids for over 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the participants were recruited from Zhujiang Hospital,Guangzhou No.12 People's Hospital,Haizhu Changgang Community,Baiyun Community Taihe Town and Tianhe Community.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
fracture | 3 years
  the participants happen to fracture

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Baiyun Community Taihe Town, Guangzhou, Guangdong
  - Guangzhou No.12 People's Hospital, Guangzhou, Guangdong
  - Haizhu Changgang Community, Guangzhou, Guangdong
  - Tianhe Community, Guangzhou, Guangdong
  - Zhujiang Hospital, Guangzhou, Guangdong